CLINICAL TRIAL: NCT03582202
Title: Organization of the Dietetic Service in a Hospital - on the Ward or Centralized?
Brief Title: Organization of the Dietetic Service in a Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-15004856
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Nutritional Disease; Malnutrition
Keywords: dietitic service, organization of service
MeSH Terms: conditions — Nutrition Disorders; Malnutrition | interventions — Nutrition Assessment; Therapeutics; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Outcomes Assessor
Masking Description: Results handled without knowledge of randomization group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietetic service (Active Comparator): Nutritional assessment and therapy by dietitian throughout the hospital stay
  Interventions: Procedure: Nutritional assessment and therapy
- standard care (Placebo Comparator): Nutritional handling by nurses supported by a dietician if needed
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Nutritional assessment and therapy — Nutritional screening, nutritional plan, follow-up and instructions on discharge
  Arms: Dietetic service
Procedure: Standard care — Nutritional handling by nurse
  Arms: standard care

SUMMARY:
In Denmark the dieticians can be organized centrally and called upon if needed, or locally in larger units, or very locally related to bed-units. The organization form is based on tradition not on measurements of quality. We wanted to compare the very local form with the traditional centralized.

Methods: Randomized, unblinded, parallel design. The intervention group (IT) was nutritionally handled by the dietician, and the control group (C) by the nurses as previously with the possibility for dietetic help from the center.

DETAILED DESCRIPTION:
All patients were screened by NRS-2002 and had their estimated needs calculated (equations in IT, tables in C). The IT was in addition assessed for adapted weight-loss, counseled with a plan for nutrition and followed-up daily by the dietician if at nutritional risk. All patients were re-screened weekly and had their intake registered. Hand-grib-strength (HGS) was measured in both groups at admittance and discharge, and weight three times weekly.

The primary endpoint was re-admission rate to hospital within 2 months.

ELIGIBILITY:
Inclusion Criteria:

* adult
* acutely admitted to hospital

Exclusion Criteria:

* dementia
* unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04-18 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
re-admission-rate after discharge (%) | 2 months
  admission for the same diagnosis

SECONDARY OUTCOMES:
intake of protein during hospital stay | 1 week
  % of estimated needs
intake of energy during hospital stay | 1 week
  % of estimated needs

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No